CLINICAL TRIAL: NCT04249908
Title: A Non-randomized, Open, Single-dose, Parallel Designed Clinical Study to Evaluate Safety and Pharmacokinetic Characteristics After Oral Administration of Besivo® in Patients With Renal Impairment and Healthy Adult Volunteers
Brief Title: Pharmacokinetics of Besifovir in Adults With Normal and Impaired Renal Function
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID-BVCL-103
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Subjects (Active Comparator)
  Interventions: Drug: Besifovir Dipivoxil Maleate
- Mild Renal Impairment (RI) (Experimental)
  Interventions: Drug: Besifovir Dipivoxil Maleate
- Moderate RI (Experimental)
  Interventions: Drug: Besifovir Dipivoxil Maleate
- Severe RI (Experimental)
  Interventions: Drug: Besifovir Dipivoxil Maleate

INTERVENTIONS:
Drug: Besifovir Dipivoxil Maleate — Besifovir 150 mg q.d.

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, and tolerability of a single oral dose of Besifovir and its metabolite, LB80331, in participants with normal and impaired renal function

ELIGIBILITY:
Inclusion Criteria:

All Individuals:

1. Have no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including vital signs, 12-lead electrocardiogram (ECG), or clinical laboratory tests.
2. Patients who were explained about the purpose, methods and effects of the clinical trial and then, signed a written consent form

Individuals with mild, moderate, or severe renal impairment must also meet the following additional inclusion criteria to be eligible for participation in this study:

1. Age of 19 to 65 years at the time of the screening visit.
2. A person whose body mass index (BMI) is greater than 18 kg/m^2 and less than 27 kg/m^2 at the time of the screening visit.
3. Individuals with severe renal impairment, estimated Glomerular Filtration Rate (eGFR) must be 15-29 mL/min/1.73m^2 (using the Modification of Diet in Renal Disease (MDRD) method) at the time of the screening visit.

   Individuals with moderate renal impairment, eGFR must be 30-59 mL/min/1.73m^2 (using the MDRD method) at the time of the screening visit.

   Individuals with mild renal impairment, eGFR must be 60-89 mL/min/1.73m^2 (using the MDRD method) at the time of the screening visit.
4. Stable renal impairment with no clinically significant changes within 3 months prior to the screening visit.

Individuals with normal renal function must also meet the following additional inclusion criteria to be eligible for participation in this study:

1. A healthy adult who is at least 19 years old at the time of the screening visit.
2. A person whose BMI is greater than 18 kg/m^2 and less than 30 kg/m^2 at the time of the screening visit.

Exclusion Criteria:

1. Medical history

   * Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hepatic, hematologic, neurologic, thyroid or any other medical illness or psychiatric disorder, as determined by the Investigator
   * A person with a history of chronic hepatitis B
   * A person with a history of gastrointestinal disorders (ex. Crohn's disease, ulcerative colitis, etc.) or surgery (except for simple appendectomy or herniotomy) that may affect the absorption of the investigational product.
2. A person who shows the following in the diagnostic test during the screening period.

   * Positive screening test for Hepatitis B Virus surface Antigen (HBs-Ag), human immunodeficiency virus (HIV) test, hepatitis C test, Venereal Disease Research Laboratory (VDRL) test
   * Clinically significant abnormal ECG findings.
   * Aspartate aminotransferase (AST) and aminotransferase (ALT) values exceed the upper limit of normal range (ULN) by more than 2 times.
   * Total Bilirubin, Gamma-Glutamyl Transpeptidase (γ-GTP) > 1.5 X ULN, Creatine Phosphokinase (CK) > 2 X ULN
   * Clinically significant laboratory abnormalities or abnormalities which are deemed to interfere with the ability to interpret study data.
3. A person who has a history of drug abuse or whose urine drug screening test result during the screening period came back positive for abusive drug use.
4. The contraindication of comedication drugs and diets

   * A person who has been administered with the investigational product or a bioequivalence study drug in another clinical trial within 180 days of the screening visit.
5. Other criteria

   * A woman whose urine human chorionic gonadotropin (hCG) test results were positive and who is pregnant or breastfeeding.
   * A person who has donated partial or full amount of blood within 60 days of the screening visit, who has given blood through apheresis within 28 days, or who has been transfused within 28 days.
   * History of regular alcohol intake > 21 units per week of alcohol before 28 dyas or unwilling to abstain from alcohol for study period before the start of admission until the final Completion Visit assessments.
   * A person who has smoked excessively within 28 days of the screening visit or whose (> 10 cigarettes/day) or◦ who can't quit smoking during the trial
   * Consumption of caffeine products within 28 days (caffeine drink > 7 glass/day) who can't abstain from caffeine products during the trial
   * Consumption of any grapefruit juice within 48 hours before administration of investigational product or subjects who can't abstain from grapefruit juice during the trial
   * Fertile subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 2 weeks after the administration of investigational product.
   * Unwillingness or inability to follow the procedures outlined in the protocol.
   * Subjects who are considered to be unacceptable in this study under the opinion of the investigator.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-13 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Plasma pharmacokinetics (PK) profiles of LB80331: Area under the plasma concentration-time curve (AUC)_0-t | Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72 hours
  This endpoint will measure the plasma PK profiles of LB80331. PK parameters that will be measured include AUC_0-t
Plasma pharmacokinetics (PK) profiles of LB80331: Cmax | Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72 hours
  This endpoint will measure the plasma PK profiles of LB80331. PK parameters that will be measured include Cmax

SECONDARY OUTCOMES:
Safety profile of Besifovir as measured by incidence of adverse events and laboratory abnormalities | Up to 16 days
  Review of adverse events and safety labs

IPD SHARING:
Plan to Share IPD: No